CLINICAL TRIAL: NCT02770053
Title: Influence of Foraminal Enlargement on Postoperative Pain in Teeth With Necrotic Pulp and Apical Periodontitis: A Randomized Controlled Trial.
Brief Title: Foraminal Enlargement and Postoperative Pain.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Isparta Military Hospital (Other)
Responsible Party: Principal Investigator, Ibrahim Ethem YAYLALI, Head of Dentistry, Isparta Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IAH-2
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-05

CONDITIONS: Pain Postoperative
Keywords: Foraminal enlargement; Root canal treatment
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Endodontic treatment will be performed in teeth with necrotic pulp and periapical periodontitis. Local anaesthesia will be provided (2% Novocaine with 1:80,000 epinephrine), isolation with rubber dam and standard access cavity preparation will be done.Using 2.5 % sodium hypochlorite, canal negotiation will be done. Foraminal enlargement will be achieved with #35 K-files in foraminal enlargement group after determining working length. Coronal flaring with # 2 and #3 Gates-Glidden drills will be done. The canals will be obturated with gutta-percha and epoxy resin sealer. The treatments will be carried out in single-visit.
  Interventions: Procedure: Foraminal enlargement
- Control (Active Comparator): In the control group, no foraminal enlargement will be performed.
  Interventions: Procedure: Foraminal enlargement

INTERVENTIONS:
Procedure: Foraminal enlargement — After determining the working length, a flexible size 30 K-file will be inserted 1 mm beyond the WL and the apical foramen will be enlarged.

SUMMARY:
The purpose of this study is to determine whether enlarging the apical foramen causes postoperative pain in teeth with necrotic pulp and apical periodontitis.

DETAILED DESCRIPTION:
Foraminal enlargement (FE) is an intentional procedure that enlarges the cement canal. However, some RCTs indicate that enlarging the FE causes postoperative pain, flare-up, and destroy the apical constriction, whilst some RCTs pointed out there is no difference in terms of pain when a FE has been performed. The investigators, therefore, would like to conduct a RCT to increase both sample size and the number of published studies to do a systematic review for this topic.

ELIGIBILITY:
Inclusion Criteria:

* Mature permenent teeth having pulpal necrosis and apical periodontitis.

Exclusion Criteria:

* Systemic disorders
* Diabetes
* Pregnancy
* Less than 18 years of age
* Immunocompromised
* Patients who had taken antibiotics in the past 1 month
* Patients who had a positive history of analgesic use within the past 3 days
* Previously accessed teeth

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
4-step pain intensity measures using a Visual Analog Scale (VAS). | 7 days.
  The severity of pain in 1-7 days according to the VAS: 0-3 mild pain, 4-7 moderate pain, and 8-10 severe pain.

SECONDARY OUTCOMES:
The number of patients taking an analgesic following the endodontics treatment. | 7 days.
  The patients were asked to take an analgesic in the 7 days of time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim E YAYLALI, Ph.D., Principal Investigator — Isparta Military Hospital

IPD SHARING:
Plan to Share IPD: Yes